CLINICAL TRIAL: NCT03294226
Title: A Randomized Trial of Ambu® AuraGain™ Versus I-gel® in Young Children
Brief Title: Comparison of AuraGain With I-gel for Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical Instructor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S2017-1229
Record Dates: First submitted 2017-09-22; First posted 2017-09-26 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AuraGain (Experimental): After anesthetic induction, AuraGain is inserted for airway management. Size of the device is selected according to the manufacturer's recommendation; size 1.5 for 5-10kg, size 2 for 10-20kg.
  Interventions: Device: AuraGain
- I-gel (Active Comparator): After anesthetic induction, I-gel is inserted for airway management. Size of the device is selected according to the patient's weight; size 1.5 for 5-10kg, size 2 for 10-20kg.
  Interventions: Device: I-gel

INTERVENTIONS:
Device: AuraGain — After anesthetic induction without neuromuscular blocking agent, AuraGain is inserted.
  Arms: AuraGain
Device: I-gel — After anesthetic induction without neuromuscular blocking agent, I-gel is inserted.
  Arms: I-gel

SUMMARY:
Children from 6 months to 6 years are randomly allocated into AuraGain group or I-gel group. After anesthetic induction without neuromuscular blocking agent, assigned device in inserted by skillful anesthesiologist. The outcome measures are recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status: 1-3
* age: from 6 months to 6 year
* body weight: 5-20kg
* patients undergoing upper/lower extremity surgery at supine position

Exclusion Criteria:

* patients who do not want to participate in this study
* patients with known difficult airway including congenital facial anomaly or history of difficult airway management
* patients with aspiration risk (gastrointestinal stenosis or stricture)
* patients with symptom of upper respiratory infection on the day of surgery
* patients scheduled for day surgery
* patients judged as not eligible by researchers for other reasons

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-24 (Actual)

PRIMARY OUTCOMES:
requirement of additional airway maneuver | during placement/maintenance of the device
  including adjustment of head/neck position or insertion depth and taping of the device

SECONDARY OUTCOMES:
insertion time | during placement of the device
success rate | during placement of the device
ease of gastric tube insertion | within 10 minutes after device insertion
adverse effect at operating room | during anesthesia
  aspiration of gastric fluid, hypoxia, SpO2<90%, bronchospasm, dental/tongue/lip trauma, staining of blood on the removed device
postoperative adverse effect | within postoperative 24 hours
  sore throat, hoarseness, airway obstruction
fiberoptic view of glottis | within 10 minutes after device insertion
  Brimacombe score
oropharyngeal leak pressure | at 1 minute after device insertion, at 10 minutes after device insertion

CONTACTS AND LOCATIONS:
Overall Officials: Won Uk Koh, M.D., Ph.D., Principal Investigator — University of Ulsan, College of Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided